CLINICAL TRIAL: NCT05184621
Title: The Effectiveness and Safety of Low-intensity Single-wavelength Red Light in Controlling High Myopia in Children and Adolescents：A Randomized, Controlled, Multicenter Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Zuoguan Medical Equipment Co., Ltd. at Suzhou Industrial Park (Unknown); Children's Hospital of Soochow University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai East Hospital (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Shanxi Eye Hospital (Other)
Responsible Party: Principal Investigator, XuYan, Deputy Chief Doctors, Shanghai Eye Disease Prevention and Treatment Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ShanghaiEye
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Age 3 to 16 Years (Inclusive), Male or Female; Clinical Diagnosis Confirming That Myopia Has Occurred in at Least One Eye; The Guardian Voluntarily Signed the Subject's Informed Consent Form
Keywords: high myopia; red light; children and adolescents

STUDY DESIGN:
Intervention Model Description: Main efficacy indicators. Axial length changes in the left and right eyes (30± 14 days, 90± 14 days, 180± 14 days, 270± 14 days, and 365± 14 days).Secondary efficacy indicator: change in equivalent spherical lens after astigmatism (day 365±14)
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- efficacy (Active Comparator): Including Primary outcome: changes in axial length of the eye. Secondary outcome: Equivalent spherical lens variation Other indicators: ① Changes in visual acuity with lenses, corrected visual acuity, and intraocular pressure.② Observation of changes in corneal thickness, anterior chamber depth, ciliary body thickness, and crystal thickness.Observation of fundus tissue structure of macula and peri-optic disc area. Observation of fundus choroidal/retinal thickness.Adherence index: frequency of device use.
  Interventions: Other: Eyesing Redlight Instrument
- safety (Active Comparator): Description of safety parameters: Adverse events, device defects during the test.
  Method and time selection for evaluation, recording, and analysis of safety parameters. Adverse events and device defects were recorded from the beginning of each subject's enrollment to the end of the group for evaluation. Safety indicators:① Incidence of allergic reactions.② Posterior image time more than 5 minutes.③ The decrease of near vision.④ The grade of side effects such as self-induced photophobia and blurred vision.⑤ Elevated intraocular pressure, headache, nausea, and vomiting, etc.
  Interventions: Other: Eyesing Redlight Instrument

INTERVENTIONS:
Other: Eyesing Redlight Instrument — Eyesing Instrument developed by Suzhou Industrial Park Zoguan Medical Equipment Co. and conventional optometry.

SUMMARY:
Objective: To study the effectiveness and safety of low-intensity single wavelength red light in controlling high myopia in children and adolescents.

Methods: Subject population: Children aged 3-16 years who have high myopia. Sample size: 190 subjects were planned to be enrolled and assigned to the test or control group in a 1:1 ratio.

DETAILED DESCRIPTION:
Design: The trial was a randomized, controlled, multicenter clinical trial. A total of 190 children aged 3-16 years with high myopia were selected and divided into 95 cases in the test group and 95 cases in the control group. The test group was treated with the Eyesing Instrument developed by Suzhou Industrial Park Zoguan Medical Equipment Co. and conventional optometry. The safety and efficacy of the low-energy laser device in the test group were evaluated by comparing the changes in myopia between the two groups during the observation period. Subjects were screened after signing the informed consent form (performed as early as 7 days before the randomization), and the examination used for screening could use the results of eye examinations performed within 1 week at our hospital, and they were enrolled after confirming that they met the inclusion criteria. On the same day, the grouping was done by randomization, and the glasses were prescribed or the glasses were prescribed in combination with the device according to the grouping results. Visits were performed at 30± 14 days, 90± 14 days, 180± 14 days, 270± 14 days, and 365± 14 days

ELIGIBILITY:
Inclusion Criteria:

1. age 3 to 16 years (inclusive), male or female
2. clinical diagnosis confirming that myopia has occurred in at least one eye.
3. the guardian voluntarily signed the "Subject's Informed Consent Form"

   Exclusion Criteria:
   * history of photosensitivity, glaucoma, glaucoma syndrome, high intraocular pressure, macular lesion or injury in the fundus ② corneal curvature examination, the average K value of the anterior surface of the cornea ≥ 45; ③ combined with heart, liver, kidney and other systemic diseases and prior.

     * Combination of cardiac, hepatic, renal, and other systemic diseases and congenital myopia; ④ Combination of ocular trauma and congenital myopia.

       ④ Combined with ocular trauma and chronic ocular diseases such as apparently oblique or operated eyes, atopic keratoconjunctivitis, etc.; ⑤ Previous presence of entropion.

       ⑤ Those with previous entropion and other eye diseases such as severe corneal and conjunctival infections; ⑥ Those with combined neurological diseases and other eye diseases.

       (6) Those with combined neurological disorders and allergies or contraindications to atropine drugs or other therapeutic drugs; (7) Albinism and psoriasis.

       (7) Patients with albinism, psoriasis, nephrotic syndrome, systemic lupus erythematosus, diabetes mellitus, and other immune system and systemic diseases; (8) Epilepsy, psychiatric disorders.

       ⑧ epilepsy, mental disorders who cannot communicate normally.
       * Previously treated with other treatments to control the development of myopia such as anticholinergic drugs such as atropine within 3 months, or involved in other functional
       * Previously treated with other treatments to control the development of myopia, such as anticholinergic drugs like atropine within 3 months, or involved in other studies related to functional frame lenses, multifocal soft lenses, etc.

   Other conditions judged by the investigator to be unsuitable for participation in the study

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Axial length changes | 30± 14 days, 90± 14 days, 180± 14 days, 270± 14 days, and 365± 14 days
  Axial length changes in the left and right eyes

SECONDARY OUTCOMES:
change in equivalent spherical | day 365±14
  change in equivalent spherical in both eyes

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Zou, advanced, Principal Investigator — Shanghai Genral Hospital/Shanghai Eye disease Treatment&Prevention Center
Locations (1):
- Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] He M, Zeng J, Liu Y, Xu J, Pokharel GP, Ellwein LB. Refractive error and visual impairment in urban children in southern china. Invest Ophthalmol Vis Sci. 2004 Mar;45(3):793-9. doi: 10.1167/iovs.03-1051. PMID 14985292
- [Result] Zhao J, Pan X, Sui R, Munoz SR, Sperduto RD, Ellwein LB. Refractive Error Study in Children: results from Shunyi District, China. Am J Ophthalmol. 2000 Apr;129(4):427-35. doi: 10.1016/s0002-9394(99)00452-3. PMID 10764849
- [Result] Maul E, Barroso S, Munoz SR, Sperduto RD, Ellwein LB. Refractive Error Study in Children: results from La Florida, Chile. Am J Ophthalmol. 2000 Apr;129(4):445-54. doi: 10.1016/s0002-9394(99)00454-7. PMID 10764851
- [Result] Pokharel GP, Negrel AD, Munoz SR, Ellwein LB. Refractive Error Study in Children: results from Mechi Zone, Nepal. Am J Ophthalmol. 2000 Apr;129(4):436-44. doi: 10.1016/s0002-9394(99)00453-5. PMID 10764850
- [Derived] Xu Y, Cui L, Kong M, Li Q, Feng X, Feng K, Zhu H, Cui H, Shi C, Zhang J, Zou H. Repeated Low-Level Red Light Therapy for Myopia Control in High Myopia Children and Adolescents: A Randomized Clinical Trial. Ophthalmology. 2024 Nov;131(11):1314-1323. doi: 10.1016/j.ophtha.2024.05.023. Epub 2024 Jun 6. PMID 38849054

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT05184621/Prot_SAP_002.pdf
  • Informed Consent Form (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT05184621/ICF_001.pdf